CLINICAL TRIAL: NCT04991220
Title: Evaluation of the Changes of Pleth Variability Index During Preoxygenation for Predicting Hypotension During Induction of Anesthesia in Surgical Patients; Prospective Observational Study
Brief Title: Evaluation of the Changes of Pleth Variability Index During Preoxygenation for Predicting Hypotension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: GEMSKOREA (Unknown)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2106-029-1232
Record Dates: First submitted 2021-07-23; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Hypotension on Induction
Keywords: Hypovolemia; Pulse Wave Analysis; Hypotension; Anesthesia, General
MeSH Terms: conditions — Hypovolemia; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- preoxygenation (Experimental): Taking 8 deep breaths at 10 l/min of 100% oxygen for 1 minute with forced inspiration for pre-oxygenation
  Interventions: Procedure: Preoxygenation

INTERVENTIONS:
Procedure: Preoxygenation — Taking 8 deep breaths at 10 l/min of 100% oxygen for 1 minute with forced inspiration for pre-oxygenation

SUMMARY:
The aim of this study is to investigate whether the change in pleth variation index (PVI) according to preoxygenation can predict hypotension during anesthesia induction.

DETAILED DESCRIPTION:
In patients with hypovolemia or dehydration, pulse pressure variation can be increased by spontaneous forced inspiratory breathing. PVI is a noninvasive method of indicator of fluid responsiveness like purse pressure variation. We expected that the amount of change in PVI between at the time of entering operating room and after preoxygenation with forced inspiration method could be different depending on the patient's volume status.

After entering operating room, monitoring devices, anesthesia depth sensor, and Radical-7® Pulse CO-Oximeter® are attached. Patients rest for 5 minutes, and then baseline systolic blood pressure, diastolic blood pressure, mean blood pressure, and heart rate are collected every 1-minute. Pleth variability index (PVI), perfusion index (PI) are also measured continuously. For pre-oxygenation of anesthesia, take 8 deep breaths at flow 10 l/min of 100% oxygen for 1 minute with maximally forced inspiration. After that, for 2 minutes, patients breathe as usual while maintaining oxygen supply. until tracheal intubation or laryngeal mask insertion. Anesthesia is induced with target concentration infusion of 4.0 ng/ml of remifentanil and 4.0 ug/ml of propofol. When the patient loses consciousness, rocuronium 1.0 mg/kg is administrated and endotracheal tube or laryngeal mask is inserted 2 minutes after. PVI, PI, blood pressure, and heart rate are measured until tracheal intubation or laryngeal mask insertion. Anesthesia induction-related hypotension is defined as a decrease in mean arterial pressure below 60 mmHg at any timepoint from baseline parameter collection to until airway device insertion. The parameters are analyzed by comparing between groups with and without anesthesia induction-related hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective surgery under general anesthesia

Exclusion Criteria:

* (1) American Society of Anesthesiologists (ASA) physical status classification III or higher (2) Patients with cognitive impairment who are unable to follow instructions (3) Patients with pulmonary dysfunction (4) Other patients who are judged inappropriate to the experiment by the researcher

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-08-30 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Hypotension during anesthesia induction | from start of anesthesia induction to just before intubation
  When mean blood pressure decreases to less than 60 mmHg at least once from the administration of anesthetic agent to just before intubation

SECONDARY OUTCOMES:
Systolic blood pressure | from entering operating room to just before intubation
  systolic blood pressure with non-invasive blood pressure at 1-minute intervals.
Diastolic blood pressure | from entering operating room to just before intubation
  diastolic blood pressure with non-invasive blood pressure at 1-minute intervals.
Heart rate | from entering operating room to just before intubation
  heart rate which was measured continuously.
Perfusion index | from entering operating room to just before intubation
  Perfusion index from Radical-7® Pulse CO-Oximeter® which was measured continously.
Pulse oximetry plethysmographic waveform; ΔPOP | from the administration of anesthetic agent to just before intubation
  Respiratory variations in the pulse oximetry plethysmographic waveform amplitude
Pleth Variability Index (PVi®) | from entering operating room to just before intubation
  the relative variability of the pleth waveform (perfusion index) detected from a Radical-7® Pulse CO-Oximeter®
Saturation of percutaneous oxygen | from entering operating room to just before intubation
  from a Radical-7® Pulse CO-Oximeter®

CONTACTS AND LOCATIONS:
Overall Officials: Hee Soo Kim, M.D., PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Billard V, Moulla F, Bourgain JL, Megnigbeto A, Stanski DR. Hemodynamic response to induction and intubation. Propofol/fentanyl interaction. Anesthesiology. 1994 Dec;81(6):1384-93. doi: 10.1097/00000542-199412000-00013. PMID 7992907
- [Background] Tsuchiya M, Yamada T, Asada A. Pleth variability index predicts hypotension during anesthesia induction. Acta Anaesthesiol Scand. 2010 May;54(5):596-602. doi: 10.1111/j.1399-6576.2010.02225.x. Epub 2010 Mar 10. PMID 20236098
- [Background] Hug CC Jr, McLeskey CH, Nahrwold ML, Roizen MF, Stanley TH, Thisted RA, Walawander CA, White PF, Apfelbaum JL, Grasela TH, et al. Hemodynamic effects of propofol: data from over 25,000 patients. Anesth Analg. 1993 Oct;77(4 Suppl):S21-9. PMID 8214693
- [Background] Berthoud M, Read DH, Norman J. Pre-oxygenation--how long? Anaesthesia. 1983 Feb;38(2):96-102. doi: 10.1111/j.1365-2044.1983.tb13925.x. PMID 6402951
- [Background] Baraka AS, Taha SK, Aouad MT, El-Khatib MF, Kawkabani NI. Preoxygenation: comparison of maximal breathing and tidal volume breathing techniques. Anesthesiology. 1999 Sep;91(3):612-6. doi: 10.1097/00000542-199909000-00009. PMID 10485768
- [Background] Bagci S, Muller N, Muller A, Heydweiller A, Bartmann P, Franz AR. A pilot study of the pleth variability index as an indicator of volume-responsive hypotension in newborn infants during surgery. J Anesth. 2013 Apr;27(2):192-8. doi: 10.1007/s00540-012-1511-6. Epub 2012 Nov 7. PMID 23132180
- [Background] Chu H, Wang Y, Sun Y, Wang G. Accuracy of pleth variability index to predict fluid responsiveness in mechanically ventilated patients: a systematic review and meta-analysis. J Clin Monit Comput. 2016 Jun;30(3):265-74. doi: 10.1007/s10877-015-9742-3. Epub 2015 Aug 5. PMID 26242233
- [Background] Wu Y, Zhang F, Sun K, Yu L, Zhang H, Yan M. [Evaluation of pleth variability index for predicting hypotension during induction of anesthesia in surgical patients]. Zhonghua Yi Xue Za Zhi. 2014 Nov 4;94(40):3167-70. Chinese. PMID 25573314
- [Background] Larsen SL, Lyngeraa TS, Maschmann CP, Van Lieshout JJ, Pott FC. Cardiovascular consequence of reclining vs. sitting beach-chair body position for induction of anesthesia. Front Physiol. 2014 May 19;5:187. doi: 10.3389/fphys.2014.00187. eCollection 2014. PMID 24904427
- [Background] Kusumoto FM, Schoenfeld MH, Barrett C, Edgerton JR, Ellenbogen KA, Gold MR, Goldschlager NF, Hamilton RM, Joglar JA, Kim RJ, Lee R, Marine JE, McLeod CJ, Oken KR, Patton KK, Pellegrini CN, Selzman KA, Thompson A, Varosy PD. 2018 ACC/AHA/HRS Guideline on the Evaluation and Management of Patients With Bradycardia and Cardiac Conduction Delay: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2019 Aug 20;74(7):e51-e156. doi: 10.1016/j.jacc.2018.10.044. Epub 2018 Nov 6. No abstract available. PMID 30412709
- [Background] Reich DL, Bennett-Guerrero E, Bodian CA, Hossain S, Winfree W, Krol M. Intraoperative tachycardia and hypertension are independently associated with adverse outcome in noncardiac surgery of long duration. Anesth Analg. 2002 Aug;95(2):273-7, table of contents. doi: 10.1097/00000539-200208000-00003. PMID 12145033
- [Background] Sheldon RS, Grubb BP 2nd, Olshansky B, Shen WK, Calkins H, Brignole M, Raj SR, Krahn AD, Morillo CA, Stewart JM, Sutton R, Sandroni P, Friday KJ, Hachul DT, Cohen MI, Lau DH, Mayuga KA, Moak JP, Sandhu RK, Kanjwal K. 2015 heart rhythm society expert consensus statement on the diagnosis and treatment of postural tachycardia syndrome, inappropriate sinus tachycardia, and vasovagal syncope. Heart Rhythm. 2015 Jun;12(6):e41-63. doi: 10.1016/j.hrthm.2015.03.029. Epub 2015 May 14. No abstract available. PMID 25980576
- [Background] Rheineck-Leyssius AT, Kalkman CJ. Influence of pulse oximeter settings on the frequency of alarms and detection of hypoxemia: Theoretical effects of artifact rejection, alarm delay, averaging, median filtering or a lower setting of the alarm limit. J Clin Monit Comput. 1998 Apr;14(3):151-6. doi: 10.1023/a:1007431305610. PMID 9676861
- [Derived] Kim YJ, Seo JH, Lee HC, Kim HS. Pleth variability index during preoxygenation could predict anesthesia-induced hypotension: A prospective, observational study. J Clin Anesth. 2023 Nov;90:111236. doi: 10.1016/j.jclinane.2023.111236. Epub 2023 Aug 26. PMID 37639751